CLINICAL TRIAL: NCT01694199
Title: A Multicenter, Randomized, Sham-Controlled, Double-Blinded Study to Evaluate the Analgesic Efficacy and Safety of Pulsed Radiofrequency Energy (PRFE) in Bunionectomy Surgery for the Treatment of Post-Operative Pain
Brief Title: Pulsed Radiofrequency Energy to Treat Post-Bunionectomy Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IDMC recommendation
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RBI.2012.003.P.2
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-01

CONDITIONS: Post-operative Pain
Keywords: Pulsed Radiofrequency Energy (PRFE); Pain; Postsurgical; Opioids; Pain relief; Medical device; Endorphins
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active study device with PRFE (Active Comparator): This study arm receives pulsed radiofrequency energy (PRFE) from an active test device.
  Interventions: Device: Pulsed Radiofrequency Energy (PRFE)
- Sham study device with no PRFE (Sham Comparator): This study arm receives no pulsed radiofrequency energy (PRFE) from a sham test device.
  Interventions: Device: No Pulsed Radiofrequency Energy (PRFE)

INTERVENTIONS:
Device: Pulsed Radiofrequency Energy (PRFE) — The intervention is pulsed radiofrequencyenergy (PRFE).
  Other Names: Provant Therapy System
  Arms: Active study device with PRFE
Device: No Pulsed Radiofrequency Energy (PRFE) — Sham (placebo) with no therapeutic device activity
  Other Names: Sham Provant Therapy System
  Arms: Sham study device with no PRFE

SUMMARY:
Multicenter, randomized, controlled, double-blind study to evaluate the use of 3 days of pulsed radiofrequency energy (PRFE) to treat pain after bunionectomy surgery.

DETAILED DESCRIPTION:
The clinical study's primary objective is to compare the overall analgesic effect of the Provant Therapy System (test device) to an identical sham device (placebo) in subjects experiencing post-operative pain following first metatarsal bunion surgery. The study hypothesis is that, over the first 72 hours (3 days) after the initial test device treatment, subjects treated with an active test device will show a statistically significant difference (reduction) in pain intensity scores when compared with subjects treated with a sham (placebo) device. Treatment with the test device will continue through the 168 hour (7 day) timepoint. Safety will be followed through 28 days.

ELIGIBILITY:
Pre-operative Inclusion Criteria:

* Adults aged 18-75 years old
* Subject is scheduled to undergo primary, unilateral first metatarsal bunionectomy (no collateral procedures) under regional/local anesthesia and sedation
* Subject meets the criteria for American Society of Anesthesiologists (ASA) Physical Status I or II.
* Subject is willing to be confined at the investigative site for approximately 4 days including the day of surgery.
* Subject is able to communicate meaningfully in English in order to complete study assessments and comply with all trial procedures.
* Willingness to give written informed consent and to comply with all parts of the study protocol.
* Female Subjects of child bearing potential are eligible only if they are not pregnant (negative pregnancy test at screening and before surgery), not lactating, and not planning to become pregnant during the study.
* Female Subjects must be post-menopausal, surgically sterile, abstinent, or practicing, or agree to practice, an effective method of birth control if they are sexually active for the duration of the study (effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier methods, and/or male partner sterilization).

Pre-Operative Exclusion Criteria:

* Subject is scheduled to undergo Base wedge osteotomy, and/or Long-Z Hart bunionectomy procedure or any other procedure that does not conform to the surgical protocol.
* Subject has received any investigational drug within 1 month prior to the Screening Visit or is enrolled in another clinical trial.
* Subject has a history of drug abuse within 5 years of the screening visit, including a history of opioid (narcotic) analgesic abuse.
* Subject has a history of any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, endocrine or psychiatric disease or disorder, or any uncontrolled medical illness that in the investigator's judgment places the Subject at unacceptable risk for surgery or receipt of investigational therapy.
* Subject has an ongoing, uncontrolled painful condition that in the opinion of the Investigator might have a confounding influence on the safety or efficacy analysis for this study.
* Subject has received systemic corticosteroid administration within 1 month prior to surgery or is scheduled to receive systemic corticosteroid therapy at any time during the course of the study.
* Subject is unwilling to abstain from alcohol from at least midnight the night before surgery through completion of all In-patient Treatment Period procedures and discharge from the investigative site.
* Subject is unwilling to refrain from smoking during his/her stay at the investigative site.
* Subject is currently receiving treatment, or has received treatment within the last two weeks, with antipsychotic drugs, monoamine oxidase inhibitors, duloxetine, gabapentin, carbamazepine, phenytoin, pregabalin or is receiving treatment with antidepressants that are not on a stable dose (the same dose for >1 month).
* Subject has a history of malignancy within the past five years with the exception of successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin and/or localized carcinoma in situ of the cervix.
* Subject has current evidence of alcohol abuse (regularly drinks more than four units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit).
* Infection (acute or chronic) involving the first metatarsal (or history of such infection) or any other disease of the foot/ankle that in the opinion of the investigator, places the Subject at increased risk for surgical complications or receipt of the investigational therapy.
* Implanted pacemaker, defibrillator, neurostimulator, bone stimulator, cochlear implant, or other implanted device with metal lead(s).
* Implanted metal in the index foot including planned intra-operative use of metallic screw or fixation device.
* History of malignancy in the treatment area.
* Subjects who are taking any dosage strength of daily opioids for more than 30 consecutive days, within the past three months prior to surgery.
* Subject with fibromyalgia, complex regional pain syndrome or other chronic pain syndromes.
* Subjects with neuropathic or sensory abnormalities of the lower extremities. Abnormal vibratory sensation and/or Semmes-Weinstein monofilament tests.
* Subject with BMI > 38.
* Subject with known hypersensitivity, intolerance or contraindication to acetaminophen, oxycodone, morphine or any agent used in the anesthetic protocol that in the opinion of the Investigator will put the Subject at increased risk.

Post-Operative Exclusion Criteria:

* The Subject does not report a score of moderate or severe on a 4-point categorical rating scale (with categories of none, mild, moderate, or severe) plus a score of ≥4 on an NPRS 11-point categorical rating scale within 8 hours after the end of surgery. End of surgery is defined as time of last suture.
* The Subject is not able to answer questions and follow commands.
* The surgical procedure from incision to closure was longer than 2 hours.
* The Subject has evidence of respiratory insufficiency, such as a respiratory rate that is less than 8 breaths per minute and arterial oxygen saturation by pulse oximetry of less than 95% with supplemental oxygen.
* There have been any significant deviations from the surgical or anesthetic protocols that would, in the opinion of the investigator, put the Subject at risk of participation in the trial, confound the analgesic endpoints of the trial or cause concern regarding the Subject's ability to participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil K. Singla, MD, Principal Investigator — Lotus Clinical Research, LLC
Locations (3):
- United States (3):
  - Lotus Clinical Research, Pasadena, California
  - Chesapeake Research Group, Pasadena, Maryland
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Study Device With PRFE | Sham Study Device With no PRFE
Started | 71 | 68
Completed | 71 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Study Device With PRFE | Sham Study Device With no PRFE | Total
Number analyzed (Participants) | 71 | 68 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 67 | 135
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (13.61) | 44.7 (13.35) | 45 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 55 | 112
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 15 | 37
  Not Hispanic or Latino | 49 | 53 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 33 | 65
  White | 38 | 28 | 66
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 71 | 68 | 139

OUTCOME MEASURES:

1. Primary Outcome: Overall Analgesic Efficacy (Via SPID 0-72 Hrs)
Description: Sum of time-weighted Pain Intensity Differences (SPID). Pain relief was assessed at completion of first treatment, 45min,60min,90min,2hrs,3hrs,4hrs,6hrs following T0 and every 2hrs between 6AM to 10PM. After 10 PM and before 6AM, pain relief assessments were done every 4hrs. Subjects rated pain relief relative to baseline using a categorical scale: 0=none; 1=a little; 2=some; 3= a lot; 4 = complete. SPIDt = ∑PID x (time(t) - time(t-1)) x PID(i). A more negative SPID value means less pain. Total score of SPID ranged from a min value of -1091550.00 in the active arm and -2120130.00 in the sham arm and a max value of 603060.00 in the active arm and 1077630.00 in the sham arm. No absolute min and max scores were calculated.
Time Frame: Treatment with the test device twice per day, over 3 days (7 total treatments)
Population: P=0.3529
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Study Device With PRFE | Sham Study Device With no PRFE
Number analyzed (Participants) | 71 | 68
units on a scale | -244890.0 [-348835.75 to -141359.18] | -258030.00 [-432672.70 to -172230.54]
Statistical Analysis 1: Comparison: Active Study Device With PRFE vs Sham Study Device With no PRFE; Test type: Superiority or Other; p = 0.3529, ANCOVA

2. Secondary Outcome: TOTPAR-Pain Relief Experienced by Patients T0-72 Hours
Description: Pain relief was assessed at completion of first study device treatment, 45 minutes, 60 minutes, 90 minutes, 2 hours, 3 hours, 4 hours, 6 hours following T0 (±5 mins). Thereafter, pain relief was assessed every 2 hours (±5 mins) between 6AM to 10PM throughout the in-patient treatment period. After 10 PM and before 6AM, pain relief assessments were done every 4 hours. Subjects rated pain relief relative to baseline pain intensity using a categorical scale: 0=none; 1=a little; 2=some; 3= a lot; 4 = complete. Based on these scores, a time weighted pain relief score was calculated, Total Pain Relief (TOTPAR). TOTPAR-Pain Relief = ∑PID x (time(t) - time(t-1)) x PID(i)."
Time Frame: Treatment with the test device twice per day, over 3 days (7 total treatments)
Measure: Geometric Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Study Device With PRFE | Sham Study Device With no PRFE
Number analyzed (Participants) | 71 | 68
units on a scale | 327974.79 [280555.32 to 375394.26] | 364873.24 [317014.18 to 412732.29]
Statistical Analysis 1: Comparison: Active Study Device With PRFE vs Sham Study Device With no PRFE; Test type: Superiority or Other; p = 0.2766, ANCOVA

3. Secondary Outcome: Opioid Consumption Measured in Morphine Equivalents T0-72 Hours
Description: The total quantity of Supplemental Opioid analgesic administered throughout the study was recorded for each Subject. Opioid consumption prior to (T0) was not considered when calculating opioid consumption endpoints.
Time Frame: Treatment with the test device twice per day, over 3 days (7 total treatments)
Measure: Median (95% Confidence Interval); unit: Morphine Equivalents
Arm/Group | Active Study Device With PRFE | Sham Study Device With no PRFE
Number analyzed (Participants) | 71 | 68
Morphine Equivalents | 23.30 [23.23 to 33.87] | 20.30 [19.21 to 27.83]
Statistical Analysis 1: Comparison: Active Study Device With PRFE vs Sham Study Device With no PRFE; P=0.1467; Test type: Superiority or Other; p = 0.1467, ANOVA

4. Secondary Outcome: Number of Participants Who Assessed Pain Control at 72 Hours as Good, Very Good, or Excellent
Description: Number of participants who assessed pain control at 72 hours as good, very good, or excellent.
Time Frame: After 3 days of treatment (T0-72 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Study Device With PRFE | Sham Study Device With no PRFE
Number analyzed (Participants) | 71 | 68
Participants | 48 | 57
Statistical Analysis 1: Comparison: Active Study Device With PRFE vs Sham Study Device With no PRFE; P = 0.5009; Test type: Superiority or Other; p = 0.5009, ANOVA

5. Secondary Outcome: Time to First Use of Supplemental Analgesic Medication
Description: The time to first supplemental analgesic use was recorded. This was defined as the time from the initiation of the first study device treatment session (T0) to the time of administration of the first dose of post-T0 supplemental medication.
Time Frame: Treatment with the test device twice per day, over 3 days (7 total treatments)
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Active Study Device With PRFE | Sham Study Device With no PRFE
Number analyzed (Participants) | 71 | 68
Minutes | 89 [70 to 99] | 87 [70 to 101]
Statistical Analysis 1: Comparison: Active Study Device With PRFE vs Sham Study Device With no PRFE; Test type: Superiority or Other; p = 0.9038, ANOVA

ADVERSE EVENTS:
Arm/Group | Active Study Device With PRFE | Sham Study Device With no PRFE
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/68
Other Adverse Events (participants affected / at risk) | 0/71 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No